CLINICAL TRIAL: NCT05534971
Title: A Randomized Study Comparing Two Techniques for Central Venous Catheter Insertion
Brief Title: Central Line Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-14157
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard technique (Active Comparator): The conventional hollow bore needle on a syringe will be used
  Interventions: Procedure: Central venous catheter insertion
- Peripheral IV (Experimental): A peripheral intravenous catheter will be used to obtain initial central venous access
  Interventions: Procedure: Central venous catheter insertion

INTERVENTIONS:
Procedure: Central venous catheter insertion — The clinical team will use the technique to establish central venous access

SUMMARY:
Two different techniques for placing a central venous catheter will be compared. The studyu team hypothesizes that clinicians randomized to the peripheral catheter technique will have higher first attempt success rates, fewer procedural complications, and a shorter mean time to procedure completion than physicians assigned to wire through hollow bore needle.

DETAILED DESCRIPTION:
Central venous catheterization (CVC) is a lifesaving procedure carried out by emergency and acute care physicians to access proximal blood vessels in order to deliver medications, blood products and other resuscitative agents. Typically, this access is achieved by threading a wire through a hollow bore needle and then placing the central venous catheter over the wire. This procedure, called the Seldinger technique, results in the cannulation of the femoral or internal jugular veins. Nowadays, physicians use concurrent ultrasound guidance rather than an anatomic landmark-based approach to increase the success rate of central venous catheterization. The wire through hollow bore needle approach requires the use of two hands to hold the needle in the vessel in order to pass a guidewire. When done under ultrasound guidance, this requires dropping the ultrasound probe in order to have both hands available to achieve vessel cannulation.

Recent research has demonstrated that cannulation of central veins can be obtained by first using a peripheral intravenous catheter rather than a hollow bore needle. This technique requires just one hand, thereby allowing the physician to continue use of the ultrasound. Furthermore, the peripheral intravenous catheter is more stable within the vein than the hollow bore needle and less likely than the needle to damage the vessel wall when the catheter is jiggled. This is the same technique used to place mid-lines, a hybrid technique that incorporates the Seldinger technique and a peripheral intravenous catheter.

ELIGIBILITY:
Inclusion Criteria:

Adult patients in the emergency department who require ultrasound guided central line placement are eligible for participation and will be referred for participation in the study by the clinical team.

Exclusion Criteria:

* Inherited, acquired, or medication related coagulopathy or thrombocytopenia (platelets < 100,000). Patients will not be excluded for use of aspirin or other anti-platelet medication.
* Previous central venous access at the same anatomical site.
* Any indwelling catheter or wire that could potentially interfere with central line placement
* Anterior border of the target vein deeper than 3.5cm

Or for any clinical feature that would interfere with obtaining informed consent including dementia, delirium, or encephalopathy, as determined by the clinical attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Only 1 attempt | 20 minutes
  The frequency with which the central line can be placed with only one attempt will be summarized. Each attempt is defined by skin penetration

SECONDARY OUTCOMES:
Unable to place central line | 20 minutes
  The frequency with which the clinical team is unable to place the central line at that clinical site using the assigned technique will be summarized by study arm.
Number of attempts | 20 minutes
  Total number of required attempts (skin penetration) will be summarized by study arm.
Number of attempted guidewire passages | 20 minutes
  Total number of attempted guidewire passages, defined as the number of times a guidewire must be attempted to be passed, will be determined. Results will be summarized by study arm.
Time taken for completion of the procedure | 20 minutes
  The duration of time from skin penetration to wire out will be summarized by study arm using basic descriptive statistics.
Procedure-related adverse events | 20 minutes
  Procedure related adverse events including pneumothorax, incorrect vessel cannulation, and bleeding requiring application of pressure will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No